CLINICAL TRIAL: NCT01765751
Title: Cervical Distraction Minimal Intervention Development: Translating From Basic to Clinical Studies
Brief Title: Manual Cervical Distraction: Measuring Chiropractic Delivery for Neck Pain Clinical Trial
Acronym: MCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: U19AT004663 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2013-01-10 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Neck Pain; Pain in Arm, Unspecified
Keywords: Cervical pain; Neck pain; Arm pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Manual Cervical Distraction High Force (Active Comparator): Manual Cervical Distraction forces will be limited to greater than 50N in the high force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
  Interventions: Procedure: Manual Cervical Distraction
- Manual Cervical Distraction Medium Force (Active Comparator): Manual Cervical Distraction forces will be limited to between 20N-50N in the medium force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
  Interventions: Procedure: Manual Cervical Distraction
- Manual Cervical Distraction Low Force (Sham Comparator): Manual Cervical Distraction forces will be limited to less than 20N in the low force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
  Interventions: Procedure: Manual Cervical Distraction

INTERVENTIONS:
Procedure: Manual Cervical Distraction — Manual Cervical Distraction (MCD) is a form of Low Velocity Variable Amplitude Spinal Manipulation (LVVA-SM). MCD procedure is performed with participant lying prone on a load instrumented table with moveable headpiece allowing guided head movement while recumbent. Clinician gently grasps posterior aspect of participant's neck with a broad contact (contact hand) between thumb and index finger at specific vertebral level. With opposite hand, clinician grasps control handle. Using contact hand, clinician exhibits superior traction to maintain a contact at a single vertebral level and ensuring a gentle movement via contact with control handle. Goal is to create a slow rhythmic (1-3 sec) localized distractive movement. In this trial, only axial distraction (Cox protocol 1) will be used.

SUMMARY:
The purpose of the Manual Cervical Distraction: Measuring Chiropractic Delivery for Neck Pain Clinical Trial is to examine the patient-centered clinical and biomechanical outcomes, doctor treatment delivery, and believability characteristics of a commonly used chiropractic procedure for the treatment of neck- or neck-related arm pain or disability.

DETAILED DESCRIPTION:
The purpose of the Manual Cervical Distraction (MCD): Measuring Chiropractic Delivery for Neck Pain Clinical Trial is to examine the patient-centered clinical and biomechanical outcomes, and believability characteristics of a manually-localized cervical distraction procedure for the treatment of neck- or neck-related arm pain or disability. One challenging issue in the study of manual therapies, including spinal manipulation (SM), is the development of sham and/or minimal intervention procedures suitable for use with control groups in clinical trials. With SM, active treatment requires substantial physical contact between a study clinician and the study participant, either directly or through a mechanical intermediary. Consequently, it is difficult to introduce differences in manual therapy procedures that distinguish sham and/or minimal interventions from the active treatment, but are not immediately obvious to the study participant. Another challenging issue is training clinicians to deliver a standardized SM treatment within specified force ranges. The muscles surrounding the neck could alter the forces transmitted to the cervical spine, and could alter the treatment effectiveness. The purpose of this pilot randomized controlled trial is to examine the patient-centered clinical, biomechanical, and believability outcome characteristics of a manually-localized cervical distraction procedure for the treatment of neck or neck-related arm pain or disability. We also will evaluate the ability of the doctor of chiropractic to deliver the MCD treatment within specified force ranges. An exploratory aim of this study is to evaluate EMG measurement during MCD delivery.

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 70 years (inclusive).
* Mechanical neck pain or neck-related upper extremity pain lasting at least 4 weeks duration.
* Mechanical neck pain or neck-related upper extremity pain classified as Quebec Task Force (QTF) 2-4.
* Naïve to flexion-distraction manual therapy procedures to cervical area.
* Average neck pain in the past 24 hours rated between 3 and 7 on a 0-10 Pain Numerical Rating Scale (NRS) at Phone Screen and Baseline 1 Interview.
* Signed Informed Consent Document.

Exclusion Criteria

* Doctor of chiropractic or current or former chiropractic student.
* Average neck pain in past 24 hours rated 0-2 or 8-10 on a 0-10 Pain NRS at Phone Screen and Baseline 1 Interview.
* Neck pain from other than somatic tissues as determined by history and clinical examination.
* Surgery to cervical-thoracic area within the past 6 months.
* Recent fracture in the cervico-thoracic spine or ribs within the past 8 weeks.
* Injections for pain in neck, shoulders, arms or hands in the past 4 weeks.
* Neck pain classified as QTF 1, 5-11.
* Unwillingness to postpone use of all types of manual treatment for neck pain, except those provided in the study for the duration of the study.
* Inability or unwillingness to comply with study protocols.
* Bone or joint pathologies representing a contraindication to study procedures.
* Any single or multisegmental fusion (surgical or congenital) of the 1st through the 7th cervical vertebrae.
* Other safety concerns as determined by the clinical evaluation/opinion at case review.
* Unable to tolerate study procedures.
* Uncontrolled hypertension: systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg.
* Simultaneous clinical management for a health condition that compromises ability to deliver study treatment or assess health status.
* Inability to read or verbally comprehend English.
* Drug or alcohol abuse or dependence, suspected or confirmed through self-report questionnaires and clinical interview.
* Depression rated as ≥ 29 on the Beck Depression Inventory.
* Cognitive or memory impairment identified during eligibility exam.
* Pregnancy, under either of the following 2 circumstances: 1) Participant safety, if participant is unable to tolerate or undergo study procedures; or 2) Fetus safety, if x-rays are required for diagnosis.
* Weight greater than 300 lbs (table weight limit).
* Referral for evaluation, diagnosis, or management of other health conditions, or additional diagnostics required for neck pain diagnosis.
* Retention of legal advice or seeking a health-related insurance claim.
* Household member previously enrolled in MCD Clinical Trial.
* Compliance concerns identified during baseline eligibility process.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maruti R. Gudavalli, PhD, Principal Investigator — Palmer College of Chiropractic
Locations (1):
- Palmer Center for Chiropractic Research, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the resulting manuscripts have been published, data sets will be provided for public access. Potential investigators can contact one of the Co-PIs to present their hypothesis, study design, instruments and/or data on which to focus, and resources required. Depending upon the needs and desires of the requesting party, the data that are shared may include analytic tables or de-identified or limited data sets that are transmitted to the requesting parties for additional analyses.

REFERENCES:
- [Background] Gudavalli MR, Vining RD, Salsbury SA, Goertz CM. Training and certification of doctors of chiropractic in delivering manual cervical traction forces: Results of a longitudinal observational study. J Chiropr Educ. 2014 Oct;28(2):130-8. doi: 10.7899/JCE-14-18. Epub 2014 Sep 19. PMID 25237767
- [Background] Vining RD, Salsbury SA, Pohlman KA. Eligibility determination for clinical trials: development of a case review process at a chiropractic research center. Trials. 2014 Oct 24;15:406. doi: 10.1186/1745-6215-15-406. PMID 25344427
- [Background] Gudavalli MR, Potluri T, Carandang G, Havey RM, Voronov LI, Cox JM, Rowell RM, Kruse RA, Joachim GC, Patwardhan AG, Henderson CN, Goertz C. Intradiscal Pressure Changes during Manual Cervical Distraction: A Cadaveric Study. Evid Based Complement Alternat Med. 2013;2013:954134. doi: 10.1155/2013/954134. Epub 2013 Aug 20. PMID 24023587
- [Result] Gudavalli MR, Vining RD, Salsbury SA, Corber LG, Long CR, Patwardhan AG, Goertz CM. Clinician proficiency in delivering manual treatment for neck pain within specified force ranges. Spine J. 2015 Apr 1;15(4):570-6. doi: 10.1016/j.spinee.2014.10.016. Epub 2014 Oct 22. PMID 25452013
- [Result] Gudavalli MR, Salsbury SA, Vining RD, Long CR, Corber L, Patwardhan AG, Goertz CM. Development of an attention-touch control for manual cervical distraction: a pilot randomized clinical trial for patients with neck pain. Trials. 2015 Jun 5;16:259. doi: 10.1186/s13063-015-0770-6. PMID 26044576
- [Result] Gudavalli MR, Vining RD, Salsbury SA, Long CR, Patwardhan AG, and Goertz CM. Forces and durations measured during delivery of a manual cervical distraction procedure. Abstract presented at the World Federation of Chiropractic Conference, 2015.
- See also: Training and certification of doctors of chiropractic in delivering manual cervical traction forces: results of a longitudinal observational study. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4211585/
- See also: Eligibility determination for clinical trials: development of a case review process at a chiropractic research center. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4221721/
- See also: Intradiscal Pressure Changes during Manual Cervical Distraction: A Cadaveric Study. — https://www.ncbi.nlm.nih.gov/pubmed/24023587
- See also: Clinician proficiency in delivering manual treatment for neck pain within specified force ranges. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4375060/
- See also: Development of an attention-touch control for manual cervical distraction: a pilot randomized clinical trial for patients with neck pain. — https://www.ncbi.nlm.nih.gov/pubmed/26044576

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Cervical Distraction Low Force: Manual Cervical Distraction (MCD) forces will be limited to less than 20N in the low force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
- Manual Cervical Distraction Medium Force: Manual Cervical Distraction(MCD) forces will be limited to between 20N-50N in the medium force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
- Manual Cervical Distraction High Force: Manual Cervical Distraction (MCD) forces will be limited to greater than 50N in the high force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
Period: Overall Study
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Started | 16 | 16 | 16
Completed | 16 | 14 | 15
Not Completed | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.2) | 47.0 (11.4) | 51.2 (13.7) | 46.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 8 | 31
  Male | 5 | 4 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Range of Traction Forces
Description: We will evaluate the clinician's ability to deliver three randomly assigned manual interventions to the cervical spine within specified traction force ranges (<20 Newtons [N], 20-50N, >50N). The primary outcome of this study is to determine the accuracy and consistency of traction force delivery ranges both between clinicians and within individual clinicians. Traction force ranges (C5 contact level and Occiput contact level) will be measured at each study visit (visits 1, 2, 3, 4, 5) for 2 weeks and averaged to calculate final outcome.
Time Frame: Day 1, 4, 8, 11, 14 (Each Study Visit)
Population: *Cervical traction forces measured in Newtons (N) over four treatment visits for each participant. We recorded 23 missing values for traction forces due to 9 missing appointments (18 observations) and 5 instances of technical problems in data collection.
Measure: Mean (Standard Deviation); unit: Newtons (N)
Units Other Than Participants: Number of Observations*
Groups:
- MCD Low Force: Manual Cervical Distraction (MCD) forces will be limited to less than 20N in the low force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
- MCD Medium Force: Manual Cervical Distraction(MCD) forces will be limited to between 20N-50N in the medium force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
- MCD High Force: Manual Cervical Distraction (MCD) forces will be limited to greater than 50N in the high force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
Arm/Group | MCD Low Force | MCD Medium Force | MCD High Force
Number analyzed (Participants) | 16 | 16 | 16
Number analyzed (Number of Observations*) | 64 | 64 | 64
Newtons (N)
  C5 Contact Level: number analyzed (Number of Observations*) | 64 | 57 | 60
  C5 Contact Level | 13.82 (5.74) | 38.3 (12.12) | 65.08 (17.70)
  Occiput Contact Level: number analyzed (Number of Observations*) | 64 | 56 | 60
  Occiput Contact Level | 17.19 (4.84) | 42.87 (10.40) | 74.06 (16.08)

2. Secondary Outcome: Neck Disability Index (NDI)
Description: The NDI is a 10-item questionnaire modified from the Oswestry Low Back Pain Disability Index. The NDI has been shown to be a reliable and valid measure of disability due to neck pain, and responsive for measuring change. Study Visit 1 and Study Visit 5 Measures occur 2 weeks apart. The NDI scale is measured on a scale of 0-50, with 0 indicating no disability and 50 indicating complete disability. This measure is an adjusted mean NDI change.
Time Frame: Change from Baseline to Day 1 (Study Visit 1) and Day 14 (Study Visit 5)
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 16
units on scale | 1.3 [-1.0 to 3.5] | 4.2 [1.8 to 6.6] | 4.0 [1.8 to 6.2]
Statistical Analysis 1: Comparison: Manual Cervical Distraction Low Force vs Manual Cervical Distraction High Force; Test type: Superiority; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-0.1 to 5.6] — High vs Low group, mean difference adjusted for the baseline value of the respective variable centered at its mean. NDI also adjusted for traction-force feedback method
Statistical Analysis 2: Comparison: Manual Cervical Distraction Low Force vs Manual Cervical Distraction Medium Force; Test type: Superiority; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [0.1 to 5.9] — Medium vs Low group, mean difference adjusted for the baseline value of the respective variable centered at its mean. NDI also adjusted for traction-force feedback method
Statistical Analysis 3: Comparison: Manual Cervical Distraction Medium Force vs Manual Cervical Distraction High Force; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-3.2 to 2.7] — High vs Medium group, mean difference adjusted for the baseline value of the respective variable centered at its mean. NDI also adjusted for traction-force feedback method

3. Secondary Outcome: Neck Pain Visual Analogue Scale (VAS)
Description: The VAS has excellent metric properties, is easy to administer and score (0-100mm), and is commonly used in pain research. Our anchors will be no pain (score of 0) to worst pain imaginable (score of 100). We will ask participants to rate their current neck pain at baseline and pre-/post-treatment for all 5 study visits. This measure is adjusted mean neck pain VAS change. A single value was calculated by averaging.
Time Frame: Change from Baseline, Day 1, 4, 8, 11, 14 (Pre- and Post-Study Visits 1, 2, 3, 4, 5)
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 16
mm | 9.1 [-1.6 to 19.8] | 18.9 [7.7 to 30.1] | 24.7 [13.9 to 35.5]
Statistical Analysis 1: Comparison: Manual Cervical Distraction Low Force vs Manual Cervical Distraction High Force; Test type: Superiority; Mean Difference (Final Values) = 15.6, 95% CI 2-sided [1.6 to 29.7] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Manual Cervical Distraction Low Force vs Manual Cervical Distraction Medium Force; Test type: Superiority; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [-3.7 to 23.3] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Manual Cervical Distraction Medium Force vs Manual Cervical Distraction High Force; Test type: Superiority; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-8.6 to 20.3] — [estimate comment as in outcome 2, analysis 3]

4. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS-43)
Description: The PROMIS-43 questionnaire will be used to measure general functional health status. PROMIS-43 questions measure physical function, anxiety, depression, fatigue, sleep disturbance, social role satisfaction, and pain interference and intensity.
  The table below displays the mean score at baseline. On the T-score metric & interpretation:
  * A score of 40 is one SD lower than the mean of the reference population (REF POP).
  * A score of 60 is one SD higher than the mean of the REF POP.
  * For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus a score of 60 is one SD above the average REF POP. This could be a desirable or undesirable outcome, depending upon the concept being measured. For Physical Function and Satisfaction with Social Role, higher scores reflect a better outcome, while for the remaining concepts, higher scores reflect a worse outcome.
  PROMIS - Pain Interference adjusted for baseline neck pain VAS.
Time Frame: Change from Baseline to Day 14 (Study Visit 5)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | MCD Low Force | MCD Medium Force | MCD High Force
Number analyzed (Participants) | 16 | 16 | 16
T-score
  PROMIS - Pain Interference (baseline) | 53.2 (6.7) | 54.9 (5.2) | 51.2 (5.6)
  PROMIS - Pain Interference (Day 14) | 50.0 (8.4) | 49.6 (7.5) | 51.6 (4.9)
  PROMIS - Physical Function (baseline) | 27.7 (5.2) | 25.3 (5.0) | 26.4 (4.5)
  PROMIS - Physical Function (Day 14) | 27.2 (6.3) | 25.7 (4.8) | 25.8 (3.7)
  PROMIS - Fatigue (baseline) | 50.4 (10.9) | 46.4 (9.3) | 47.1 (7.2)
  PROMIS - Fatigue (Day 14) | 53.8 (12.6) | 47.0 (6.4) | 45.6 (7.4)
  PROMIS - Sleep Disturbance (baseline) | 51.3 (3.0) | 51.3 (3.0) | 51.5 (2.6)
  PROMIS - Sleep Disturbance (Day 14) | 51.2 (2.6) | 52.6 (4.1) | 49.8 (2.4)
  PROMIS - Anxiety (baseline) | 46.8 (10.9) | 47.5 (8.0) | 45.3 (8.4)
  PROMIS - Anxiety (Day 14) | 45.3 (9.8) | 46.2 (7.2) | 43.4 (5.8)
  PROMIS - Depression (baseline) | 42.6 (6.8) | 43.9 (7.8) | 43.6 (5.5)
  PROMIS - Depression (Day 14) | 42.8 (6.3) | 42.1 (5.6) | 40.4 (4.6)
  PROMIS - Satisfaction with Social Role (baseline) | 51.7 (8.5) | 53.6 (7.6) | 54.3 (6.5)
  PROMIS - Satisfaction with Social Role (Day 14) | 50.9 (11.2) | 55.2 (8.0) | 53.4 (8.5)
Statistical Analysis 1: Comparison: MCD Low Force vs MCD High Force; Pain Interference; Test type: Superiority; Mean Difference (Net) = -3.9, 95% CI 2-sided [-8.1 to 0.4] — Pain Interference - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 2: Comparison: MCD Low Force vs MCD Medium Force; Pain Interference; Test type: Superiority; Mean Difference (Net) = 1.5, 95% CI 2-sided [-2.6 to 5.6] — Pain Interference - Medium vs Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 3: Comparison: MCD Medium Force vs MCD High Force; Pain Interference; Test type: Superiority; Mean Difference (Net) = -5.4, 95% CI 2-sided [-9.8 to 1.0] — Pain Interference - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 4: Comparison: MCD Low Force vs MCD High Force; Physical Function; Test type: Superiority; Mean Difference (Net) = 0.8, 95% CI 2-sided [-2.2 to 3.8] — Physical Function - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 5: Comparison: MCD Low Force vs MCD Medium Force; Physical Funtion; Test type: Superiority; Mean Difference (Net) = 0.1, 95% CI 2-sided [-2.9 to 3.2] — Physical Function - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 6: Comparison: MCD Medium Force vs MCD High Force; Physical Function; Test type: Superiority; Mean Difference (Net) = 0.7, 95% CI 2-sided [-2.4 to 3.7] — Physical Function- High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 7: Comparison: MCD Low Force vs MCD High Force; Fatigue; Test type: Superiority; Mean Difference (Net) = 5.8, 95% CI 2-sided [1.1 to 10.5] — Fatigue - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 8: Comparison: MCD Low Force vs MCD Medium Force; Fatigue; Test type: Superiority; Median Difference (Net) = 3.3, 95% CI 2-sided [-1.5 to 8.2] — Fatigue - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 9: Comparison: MCD Medium Force vs MCD High Force; Fatigue; Test type: Superiority; Mean Difference (Net) = 2.5, 95% CI 2-sided [-2.3 to 7.3] — Fatigue - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 10: Comparison: MCD Low Force vs MCD High Force; Sleep Disturbance; Test type: Superiority; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.9 to 3.5] — Sleep Disturbance - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 11: Comparison: MCD Low Force vs MCD Medium Force; Sleep Disturbance; Test type: Superiority; Mean Difference (Net) = -1.4, 95% CI 2-sided [-3.6 to 0.9] — Sleep Disturbance - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 12: Comparison: MCD Medium Force vs MCD High Force; Sleep Disturbance; Test type: Superiority; Mean Difference (Net) = 2.7, 95% CI 2-sided [0.4 to 5.0] — Sleep Disturbance - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 13: Comparison: MCD Low Force vs MCD High Force; Anxiety; Test type: Superiority; Mean Difference (Net) = -0.3, 95% CI 2-sided [-4.5 to 3.9] — Anxiety - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 14: Comparison: MCD Low Force vs MCD Medium Force; Anxiety; Test type: Superiority; Mean Difference (Net) = 1.1, 95% CI 2-sided [-2.9 to 5.1] — Anxiety - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 15: Comparison: MCD Medium Force vs MCD High Force; Anxiety; Test type: Superiority; Mean Difference (Net) = -1.4, 95% CI 2-sided [-5.7 to 2.9] — Anxiety - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 16: Comparison: MCD Low Force vs MCD High Force; Depression; Test type: Superiority; Mean Difference (Net) = -2.8, 95% CI 2-sided [-6.7 to 0.6] — Depression - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 17: Comparison: MCD Low Force vs MCD Medium Force; Depression; Test type: Superiority; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.1 to 2.6] — Depression - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 18: Comparison: MCD Medium Force vs MCD High Force; Depression; Test type: Superiority; Mean Difference (Net) = -2.0, 95% CI 2-sided [-5.4 to 1.4] — Depression - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 19: Comparison: MCD Low Force vs MCD High Force; Satisfaction with Social Role; Test type: Superiority; Mean Difference (Net) = 0.2, 95% CI 2-sided [-4.5 to 4.9] — Satisfaction with Social Role - High vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 20: Comparison: MCD Low Force vs MCD Medium Force; Satisfaction with Social Role; Test type: Superiority; Mean Difference (Net) = 3.0, 95% CI 2-sided [-1.8 to 7.7] — Satisfaction with Social Role - Medium vs. Low Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population
Statistical Analysis 21: Comparison: MCD Medium Force vs MCD High Force; Satisfaction with Social Role; Test type: Superiority; Mean Difference (Net) = -2.8, 95% CI 2-sided [-7.6 to 2.0] — Satisfaction with Social Role - High vs. Medium Group - The scale for the PROMIS measures uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population

5. Secondary Outcome: Cervical Range of Motion (cROM).
Description: Cervical ranges of motion are a measure of functional status and can be used to assess dysfunction in the cervical spine. Baseline/visit 1 ("BL") cROM is displayed for Flexion-Extension, Lateral Bending, and Rotation. The mean change in cROM from visit 1 to visit 5 ("V5 change") is also displayed.
Time Frame: Change from Day 1 (Study Visit 1) to Day 14 (Study Visit 5)
Population: The number analyzed in row differs from overall due to:
  1. Data collection issue due to equipment problems.
  2. Participants did not show up for data collection.
  3. 3 Participants were lost to follow up
Measure: Mean (Standard Deviation); unit: Degrees - Range of Motion
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 14
Degrees - Range of Motion
  BL - Mean Flexion-Extension: number analyzed (Participants) | 14 | 15 | 14
  BL - Mean Flexion-Extension | 70.2 (25.9) | 75.4 (32.4) | 78.6 (28.5)
  BL - Mean Lateral Bending | 51.6 (21.1) | 54.7 (12.1) | 49.8 (13.6)
  BL - Mean Rotation: number analyzed (Participants) | 16 | 15 | 14
  BL - Mean Rotation | 88.5 (25.4) | 91.1 (22.8) | 88.5 (19.7)
  Mean Change from BL to V5 - Flexion-Extension: number analyzed (Participants) | 13 | 11 | 13
  Mean Change from BL to V5 - Flexion-Extension | 0.8 (14.9) | 6.1 (31.7) | 4.9 (25.2)
  Mean Change from BL to V5 - Lateral Bending: number analyzed (Participants) | 15 | 12 | 13
  Mean Change from BL to V5 - Lateral Bending | -4.7 (24.3) | -2.9 (8.7) | -2.3 (24.1)
  Mean Change from BL to V5 - Rotation: number analyzed (Participants) | 15 | 12 | 14
  Mean Change from BL to V5 - Rotation | 2.3 (15.5) | -8.9 (28) | -8.1 (37.5)

6. Secondary Outcome: Procedure Believability Questionnaire
Description: We will ask all participants whether they feel the study procedure would relieve their neck pain using the Procedure Believability Questionnaire. The response choices will be: "Strongly believe the procedure will relieve my neck pain; Somewhat believe the procedure will relieve my neck pain; Somewhat believe the procedure will NOT relieve my neck pain; Strongly believe the procedure will NOT relieve my neck pain; and Don't know if the procedure will relieve my neck pain". A baseline (BL) evaluation will be completed based upon treatment description, and compared to assessments following study visit 1 (T1) and study visit 5 (T5) over a 2-week time period.
Time Frame: Baseline (BL), Day 1 (Study Visit 1/T1), Day 14 (Study Visit 5/T5)
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 16
Participants
  BL - Strongly WILL | 3 | 6 | 3
  BL - Somewhat WILL | 5 | 5 | 8
  BL - Somewhat will not | 0 | 1 | 0
  BL - Strongly will NOT | 0 | 0 | 4
  BL - Don't know | 8 | 4 | 4
  T1 - Strongly WILL | 4 | 6 | 4
  T1 - Somewhat WILL | 6 | 10 | 8
  T1 - Somewhat will not | 2 | 0 | 0
  T1 - Strongly will NOT | 1 | 0 | 1
  T1 - Don't know | 3 | 0 | 3
  T5 - Strongly WILL | 4 | 5 | 3
  T5 - Somewhat WILL | 4 | 8 | 6
  T5 - Somewhat will not | 1 | 2 | 0
  T5 - Strongly will NOT | 6 | 0 | 2
  T5 - Don't know | 1 | 0 | 3
  T5 - Missing | 0 | 1 | 2

7. Secondary Outcome: Credibility and Expectancy Questionnaire (CEQ)
Description: The CEQ is a quick and easy-to-administer questionnaire for measuring treatment expectancy and rationale credibility of interventions for use in clinical outcome studies. Participants' perceptions of the study treatments were compared across groups using the CEQ. The CEQ credibility factor relates to how logical or believable a treatment is for the patient, whereas the expectancy factor refers to the patient's beliefs about improvements that might be achieved from the treatment [61]. CEQ scores for both the credibility and expectancy factors range from 3 to 27, with higher scores indicating greater belief in treatment credibility or expectancy for clinical improvement.
Time Frame: Baseline, Day 1 (Study Visit 1), Day 14 (Study Visit 5)
Measure: Mean (Standard Deviation); unit: units on a scale (range 3-27)
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 16
units on a scale (range 3-27)
  Credibility Factor - Basline 1 Visit | 19.8 (2.2) | 23.1 (3.4) | 21.0 (3.9)
  Credibility Factor - Study Visit 1 | 15.5 (7.0) | 19.9 (5.2) | 22.1 (4.8)
  Credibility Factor - Study Visit 5 | 13.8 (8.0) | 19.9 (7.5) | 22.7 (4.0)
  Expectancy Factor - Baseline Visit 1 | 15.8 (4.0) | 19.7 (4.7) | 16.0 (6.9)
  Expectancy Factor - Study Visit 1 | 13.4 (6.2) | 17.8 (5.8) | 19.3 (6.7)
  Expectancy Factor - Study Visit 5 | 11.4 (7.8) | 15.1 (8.3) | 17.8 (6.2)

8. Other Pre Specified Outcome: Cervical Muscle Electromyographic (EMG) Activity
Description: We will describe electromyographic (EMG) activity of superficial neck muscles during delivery of the three manual interventions during visits 3 and 4. EMG measurements are an exploratory outcome variable in this study.
  RMS EMG TREATMENT DESCRIPTIONS:
  * (A) Ratio of Root Mean square (RMS) EMG during Treatment at C5/RMS EMG during maximum voluntary contraction (MVC)
  * (B) RMS EMG during Treatment at C5/RMS EMG during Prone Resting
  * (C) RMS EMG during Treatment at Occiput (OCC)/RMS EMG during MVC
  * (D) RMS EMG during Treatment at OCC/ RMS EMG during Prone Resting
  MUSCLES:
  * LES-Left erector Spinae Muscle
  * RES-Right Erector Spinae Muscle
  * LTRPS- Left Trapezius muscle
  * RTRPS- Right Trapezius Muscle
  * LSCM- Left Sternocleido Mastoid muscle
  * RSCM- Right Sternocleido Mastoid Muscle
  ACRONYM KEY:
  * RMS-Root Mean Square Value
  * MVC-Maximum Voluntary Contraction
  * C5-Cervical vertebrae contact
  * OCC-Occipital contact
  * EMG-Electromyographic activity
Time Frame: Day 8 (Study Visit 3), Day 11 (Study Visit 4)
Population: The numbers analyzed in the row differ from the overall due to: (1) Data not collected due to technical problems, (2) Patient did not show up for the visit, (3) 3 participants lost to follow up.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 13 | 15
ratio
  Visit 3 - (A) - LES: number analyzed (Participants) | 15 | 10 | 12
  Visit 3 - (A) - LES | 0.25 (0.20) | 0.26 (0.22) | 0.31 (0.25)
  Visit 3 - (A) - RES: number analyzed (Participants) | 14 | 8 | 10
  Visit 3 - (A) - RES | 0.28 (0.28) | 0.34 (0.14) | 0.16 (0.13)
  Visit 3 - (A) - LTRPS: number analyzed (Participants) | 16 | 13 | 14
  Visit 3 - (A) - LTRPS | 0.27 (0.25) | 0.23 (0.12) | 0.22 (0.20)
  Visit 3 - (A) - RTRPS: number analyzed (Participants) | 15 | 10 | 13
  Visit 3 - (A) - RTRPS | 0.42 (0.30) | 0.37 (0.26) | 0.29 (0.25)
  Visit 3 - (A) - LSCM: number analyzed (Participants) | 16 | 12 | 15
  Visit 3 - (A) - LSCM | 0.24 (0.26) | 0.22 (0.18) | 0.14 (0.10)
  Visit 3 - (A) - RSCM: number analyzed (Participants) | 16 | 11 | 15
  Visit 3 - (A) - RSCM | 0.15 (0.07) | 0.19 (0.17) | 0.13 (0.12)
  Visit 3 - (B) - LES: number analyzed (Participants) | 16 | 12 | 15
  Visit 3 - (B) - LES | 1.32 (1.04) | 2.03 (1.46) | 1.40 (0.76)
  Visit 3 - (B) - RES: number analyzed (Participants) | 15 | 12 | 11
  Visit 3 - (B) - RES | 1.67 (0.92) | 2.53 (2.12) | 2.13 (1.78)
  Visit 3 - (B) - LTRPS | 1.41 (0.44) | 1.80 (0.85) | 1.27 (0.37)
  Visit 3 - (B) - RTRPS: number analyzed (Participants) | 16 | 12 | 15
  Visit 3 - (B) - RTRPS | 1.29 (0.18) | 1.31 (0.22) | 1.20 (0.22)
  Visit 3 - (B) - LSCM: number analyzed (Participants) | 16 | 12 | 15
  Visit 3 - (B) - LSCM | 1.36 (0.50) | 1.68 (1.27) | 1.78 (1.40)
  Visit 3 - (B) - RSCM | 1.47 (0.66) | 1.83 (1.13) | 1.41 (0.66)
  Visit 3 - (C) - LES: number analyzed (Participants) | 16 | 13 | 14
  Visit 3 - (C) - LES | 0.21 (0.17) | 0.22 (0.19) | 0.25 (0.19)
  Visit 3 - (C) - RES: number analyzed (Participants) | 16 | 13 | 14
  Visit 3 - (C) - RES | 0.25 (0.22) | 0.24 (0.15) | 0.16 (0.16)
  Visit 3 - (C) - LTRPS | 0.23 (0.20) | 0.19 (0.12) | 0.24 (0.22)
  Visit 3 - (C) - RTRPS | 0.36 (0.29) | 0.36 (0.26) | 0.31 (0.29)
  Visit 3 - (C) - LSCM | 0.24 (0.24) | 0.15 (0.15) | 0.12 (0.09)
  Visit 3 - (C) - RSCM | 0.13 (0.07) | 0.17 (0.16) | 0.12 (0.08)
  Visit 3 - (D) - LES | 1.41 (0.95) | 1.54 (1.06) | 1.49 (0.88)
  Visit 3 - (D) - RES: number analyzed (Participants) | 16 | 12 | 14
  Visit 3 - (D) - RES | 1.77 (1.43) | 1.41 (0.25) | 1.58 (1.38)
  Visit 3 - (D) - LTRPS | 1.38 (0.57) | 1.47 (0.60) | 1.24 (0.19)
  Visit 3 - (D) - RTRPS | 1.68 (1.72) | 1.38 (0.28) | 1.21 (0.16)
  Visit 3 - (D) - LSCM | 1.30 (0.26) | 1.48 (0.54) | 1.69 (0.98)
  Visit 3 - (D) - RSCM | 1.32 (0.34) | 1.48 (0.43) | 1.49 (0.75)
  Visit 4 - (A) - LES: number analyzed (Participants) | 13 | 11 | 12
  Visit 4 - (A) - LES | 0.30 (0.15) | 0.25 (0.15) | 0.27 (0.19)
  Visit 4 - (A) - RES: number analyzed (Participants) | 15 | 10 | 13
  Visit 4 - (A) - RES | 0.20 (0.18) | 0.28 (0.17) | 0.20 (0.22)
  Visit 4 - (A) - LTRPS: number analyzed (Participants) | 15 | 13 | 14
  Visit 4 - (A) - LTRPS | 0.24 (0.23) | 0.22 (0.20) | 0.25 (0.24)
  Visit 4 - (A) - RTRPS: number analyzed (Participants) | 15 | 11 | 14
  Visit 4 - (A) - RTRPS | 0.43 (0.27) | 0.28 (0.22) | 0.30 (0.25)
  Visit 4 - (A) - LSCM: number analyzed (Participants) | 16 | 13 | 13
  Visit 4 - (A) - LSCM | 0.11 (0.09) | 0.27 (0.22) | 0.13 (0.09)
  Visit 4 - (A) - RSCM: number analyzed (Participants) | 16 | 12 | 13
  Visit 4 - (A) - RSCM | 0.22 (0.19) | 0.18 (0.22) | 0.15 (0.12)
  Visit 4 - (B) - LES: number analyzed (Participants) | 15 | 13 | 13
  Visit 4 - (B) - LES | 1.34 (0.83) | 1.71 (1.54) | 1.75 (1.50)
  Visit 4 - (B) - RES: number analyzed (Participants) | 15 | 12 | 14
  Visit 4 - (B) - RES | 2.17 (2.20) | 2.06 (0.92) | 1.81 (1.53)
  Visit 4 - (B) - LTRPS: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (B) - LTRPS | 1.36 (0.41) | 1.31 (0.19) | 1.84 (1.69)
  Visit 4 - (B) - RTRPS: number analyzed (Participants) | 16 | 11 | 14
  Visit 4 - (B) - RTRPS | 1.61 (1.21) | 1.14 (0.38) | 1.27 (0.13)
  Visit 4 - (B) - LSCM: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (B) - LSCM | 1.29 (0.38) | 1.82 (0.97) | 2.20 (1.29)
  Visit 4 - (B) - RSCM: number analyzed (Participants) | 16 | 12 | 13
  Visit 4 - (B) - RSCM | 1.53 (0.95) | 1.55 (1.15) | 1.67 (0.92)
  Visit 4 - (C) - LES: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (C) - LES | 0.27 (0.15) | 0.27 (0.20) | 0.22 (0.17)
  Visit 4 - (C) - RES: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (C) - RES | 0.13 (0.10) | 0.30 (0.22) | 0.15 (0.17)
  Visit 4 - (C) - LTRPS: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (C) - LTRPS | 0.23 (0.21) | 0.21 (0.20) | 0.21 (0.24)
  Visit 4 - (C) - RTRPS: number analyzed (Participants) | 16 | 12 | 14
  Visit 4 - (C) - RTRPS | 0.38 (0.27) | 0.32 (0.29) | 0.31 (0.26)
  Visit 4 - (C) - LSCM: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (C) - LSCM | 0.12 (0.15) | 0.17 (0.13) | 0.12 (0.09)
  Visit 4 - (C) - RSCM: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (C) - RSCM | 0.19 (0.17) | 0.22 (0.24) | 0.14 (0.17)
  Visit 4 - (D) - LES: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (D) - LES | 1.29 (0.54) | 1.68 (1.12) | 1.59 (1.43)
  Visit 4 - (D) - RES: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (D) - RES | 1.08 (0.51) | 1.32 (0.65) | 1.76 (1.12)
  Visit 4 - (D) - LTRPS: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (D) - LTRPS | 1.48 (0.74) | 1.40 (0.70) | 1.49 (0.56)
  Visit 4 - (D) - RTRPS: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (D) - RTRPS | 1.26 (0.50) | 1.36 (0.42) | 1.31 (0.14)
  Visit 4 - (D) - LSCM: number analyzed (Participants) | 16 | 13 | 14
  Visit 4 - (D) - LSCM | 1.65 (1.73) | 2.38 (1.86) | 2.37 (2.57)
  Visit 4 - (D) - RSCM: number analyzed (Participants) | 16 | 12 | 14
  Visit 4 - (D) - RSCM | 1.31 (0.44) | 1.54 (0.63) | 1.32 (0.40)

9. Other Pre Specified Outcome: Patient Satisfaction Questionnaire
Description: Participants' satisfaction with study procedures and staff were assessed at Study Visit 5 using standard questions. Participants rated their satisfaction with various elements of the study (e.g., treatments received, clinicians) using a 5 category response from 1 (strongly satisfied) to 5 (strongly dissatisfied) with categories collapsed into satisfied (categories 1 and 2) or not satisfied (categories 3, 4 or 5) for interpretation.
Time Frame: Day 14 (Study Visit 5)
Measure: Count of Participants; unit: Participants
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force | Manual Cervical Distraction High Force
Number analyzed (Participants) | 16 | 16 | 16
Participants
  Satisfied with Treatment | 7 | 9 | 15
  Satisfied with Clinician | 14 | 14 | 15

ADVERSE EVENTS:
Time Frame: AE data were collected during five study visits over a two week period
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of AEs may exceed the total # of people affected because some people experienced multiple AEs.
Groups:
- Manual Cervical Distraction Medium Force*: Manual Cervical Distraction(MCD) forces will be limited to between 20N-50N in the medium force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
- Manual Cervical Distraction High Force*: Manual Cervical Distraction (MCD) forces will be limited to greater than 50N in the high force group. Dosing for this clinical trial is limited to 3 sets of 5 repetitions with a hand contact on one cervical vertebra of highest clinical importance and 3 sets of 5 repetitions with a hand contact on the occiput.
Arm/Group | Manual Cervical Distraction Low Force | Manual Cervical Distraction Medium Force* | Manual Cervical Distraction High Force*
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 10/16 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Manual Cervical Distraction Low Force (N=16) | Manual Cervical Distraction Medium Force* (N=16) | Manual Cervical Distraction High Force* (N=16)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Thoracic Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck and back pain/stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Tenderness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
General soreness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache and neck/back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck, back and extremity pain/stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain/stiffness and headache and dizziness/vertigo (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain/stiffness and chest soreness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizzinesss/imbalance/vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Ear infection (Ear and labyrinth disorders) | 0 | 1 | 0
Thyroid disregulation (Endocrine disorders) | 0 | 1 | 0
Increased intraocular pressure (Eye disorders) | 0 | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory infection and joint pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes